CLINICAL TRIAL: NCT05200325
Title: Establishing Clinical Utility Evidence to Support Coverage and Reimbursement for TissueCypher®: A CPV® Randomized Controlled Trial
Brief Title: Clinical Utility Evidence for TissueCypher®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Pro00056136
Record Dates: First submitted 2021-12-09; First posted 2022-01-20 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Gastro-Intestinal Disorder; Barrett Esophagus
MeSH Terms: conditions — Digestive System Diseases; Barrett Esophagus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants, who are care providers, do not know what study arm they are included in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group does not receive educational materials about the TissueCypher diagnostic test and will treat their simulated patients with the current standard of care tools.
- Intervention Group 1 (Experimental): Intervention group 1 receives educational materials about the TissueCypher diagnostic test. These materials detail what the test does, how it is used, the validity and specifications of the test, and how to read its test report. This intervention group is then forced to use the test results in treating their simulated patients.
  Interventions: Other: Educational materials for TissueCypher
- Intervention Group 2 (Experimental): Intervention group 2 receives educational materials about the TissueCypher diagnostic test. These materials detail what the test does, how it is used, the validity and specifications of the test, and how to read its test report. This intervention group then gets to decide whether or not they want to use the TissueCypher test results for their simulated patients.
  Interventions: Other: Educational materials for TissueCypher

INTERVENTIONS:
Other: Educational materials for TissueCypher — These materials detail what the test does, how it is used, the validity and specifications of the test, and how to read its test report.
  Arms: Intervention Group 1; Intervention Group 2

SUMMARY:
Cernostics has developed a new diagnostic test, and this study will measure how gastroenterologists and foregut surgeons make diagnostic and treatment decisions when presented with different information in the context of simulated clinical cases. The results of this study could contribute to improved quality of care for patients by encouraging better care practices and adherence to evidence-based guidance. The data from this study will be provided to all participating physicians and submitted to a national journal for publication. The study plans to enroll up to 249 physicians.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified gastroenterologist or GI surgeon for at least two years
* Averages at least 20 hours per week of clinical and patient care duties over the last six months
* performs either diagnostic endoscopy, interventional endoscopy, upper GI surgery, or bariatric surgery
* practicing in the US
* english speaking
* access to the internet
* informed and voluntarily consented to be in the study

Exclusion Criteria:

* non-English speaking
* unable to access the internet
* not practicing in the US
* not averaging at least 20 hours per week of clinical or patient care duties over the last six months
* does not perform either diagnostic endoscopy, interventional endoscopy, upper GI surgery, or bariatric surgery
* does not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Clinical Performance and Value (CPV)-measured change in physician behavior | 4 months
  Change in the overall and the diagnostic and treatment evidence-based quality scores in the CPV patient simulations: difference-in-differences regression analysis between the control and the intervention groups' diagnosis and treatment of risk progression in patients with Barrett's esophagus, as measured by the participants diagnostic and treatment CPV case domain scores. In each domain of a CPV (history, physical exam, workup, diagnosis and treatment), participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum from 0 to a high potential score of up to 100 percent in each domain, where higher scores mean better outcomes.
CPV-measured evidence based management decisions | 4 months
  Evidence-based management decisions based on patient's TissueCypher® test result: Once the intervention group is exposed to the intervention, education materials on the TissueCypher (a validated diagnostic test for predicting risk progression of BE patients), the scores are measured, on a scale of 0% to 100% from round 1 (pre-exposure) to round 2 (post-exposure) and observe how the evidence-based TissueCypher results influence physicians' management decisions.
CPV-measured cost savings | 1 month
  Change in cost of BE-related care. (This cost is modeled in part by measuring differential rates of endoscopic work up/interventions/levels of care selected by each arm, and multiplying by average Medicare reimbursement rates for these workups/interventions/levels of care. The cost is also modeled by examining average per annum costs for patients suffering from BE, and multiplying by the percent of patients whose workup or therapeutic management is significantly reduced following the intervention.)

SECONDARY OUTCOMES:
CPV-measured baseline levels of variation | 4 months
  Participants completing the simulated cases, or CPVs, receive scores, on a scale from 0% to 100%, based upon the quality of care they provide. This measure will assess the baseline levels of variation in the care of pain patients among all participants, including by use case types. Baseline levels of variation will be measured in the surveillance, management and treatment of patients with Barrett's esophagus among all participants
CPV-measured use case analysis | 4 months
  Difference in the overall, and the diagnostic and treatment quality scores between control and intervention participants. Diagnostic and treatment scores are calculated as the percent correct on CPVs, and the overall score is an average score of the subcategory scores (percent correct). The score is reported on a scale from 0% to 100%. This will be examined for each of the use cases to determine in which case(s) CPV scores most improved.

CONTACTS AND LOCATIONS:
Locations (1):
- QURE Healthcare, San Francisco, California, United States

REFERENCES:
- [Derived] Peabody JW, Cruz JDC, Ganesan D, Paculdo D, Critchley-Thorne RJ, Wani S, Shaheen NJ. A Randomized Controlled Study on Clinical Adherence to Evidence-Based Guidelines in the Management of Simulated Patients With Barrett's Esophagus and the Clinical Utility of a Tissue Systems Pathology Test: Results From Q-TAB. Clin Transl Gastroenterol. 2024 Jan 1;15(1):e00644. doi: 10.14309/ctg.0000000000000644. PMID 37767993